CLINICAL TRIAL: NCT05685563
Title: Influence of Regularly Repeated Asymmetric Load on the Locomotor System in Sweep Rowers
Brief Title: Load During Sweep Rowing and the Influence on the Posture
Status: Completed | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Sponsor
Other Study IDs: Mikulík, rowing
Record Dates: First submitted 2022-12-31; First posted 2023-01-17 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Muscle Hypertonia; Postural Scoliosis; Postural; Defect
Keywords: sweep rowing; pedobarography; moiré topography; asymmetrical loading
MeSH Terms: conditions — Muscle Hypertonia | interventions — Pain Measurement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- sweep rowers: Each subject was assessed using DIERS formetic 4D and DIERS pedoscan devices. Additionally, participants in each group were assessed by FAIR test, Cluster of Laslett, trigger point palpation of the m. piriformis and Visual analogue scale.
  Interventions: Diagnostic Test: DIERS formetic 4D
- scull rowers: Each subject was assessed using DIERS formetic 4D and DIERS pedoscan devices. Additionally, participants in each group were assessed by FAIR test, Cluster of Laslett, trigger point palpation of the m. piriformis and Visual analogue scale.
  Interventions: Diagnostic Test: DIERS formetic 4D
- control non-rowers: Each subject was assessed using DIERS formetic 4D and DIERS pedoscan devices. Additionally, participants in each group were assessed by FAIR test, Cluster of Laslett, trigger point palpation of the m. piriformis and Visual analogue scale.
  Interventions: Diagnostic Test: DIERS formetic 4D

INTERVENTIONS:
Diagnostic Test: DIERS formetic 4D — Assessment of mentioned tests and their comparison.
  Other Names: trigger point palpation of the m. piriformis; DIERS pedoscan device; Visual analogue scale; FAIR test; Cluster of Laslett test

SUMMARY:
The aim is to assess the influence of asymmetric training on the locomotor system in sweep rowers. To analyse possible changes objectively, the axial position of the hull will be assessed using Moiré topography, and the symmetry of foot loading will be monitored with a pedobarograph. Furthermore, the Visual Analog scale and Cluster of Laslett will determine whether an asymmetric load can provoke pain in the lumbar region or cause a blockage in the SI joint. In the experimental study, there will be three different groups of participants. Selected sweep rowers will make the first study group. The second group will consist of scull rowers, and the last control group will consist of people with no experience with rowing. The selected participants will undergo the first measurement at the turn of the spring and summer seasons when intensive preparation for rowing competitions begins, in which sweep rowers train mainly on water and asymmetrically. The measurement results in the three groups will be further compared with each other to evaluate whether statistically significant differences can be found.

DETAILED DESCRIPTION:
Methods: 21 sweep rowers, 20 scull rowers and 23 non-rowing peers were enrolled on the study of this diploma thesis. Each subject was assessed using DIERS formetic 4D and DIERS pedoscan devices. Additionally, participants in each group were assessed by FAIR test, Cluster of Laslett, trigger point palpation of the m. piriformis and Visual analogue scale were used to assess pain intensity in the lumbar region.

ELIGIBILITY:
Inclusion Criteria for rowers:

* Training and racing exclusively in the unpaired disciplines of competitive rowing in the Czech Republic for a group of unpaired rowers
* Training and racing exclusively in the pairs disciplines of competitive rowing in the Czech Republic for the group of pairs rowers
* Dedication to rowing for more than three years
* Frequency of training at least three times a week or more

Inclusion Criteria for non-rowers:

-Engaging in sports recreationally without higher intensity training (less than three times a week) or at all.

Exclusion Criteria for rowers:

* The presence of lumbar spine pain at a time when the athlete was not yet exercising
* Presence of musculoskeletal pain caused by a condition for which the athlete is actively being treated (Morbus Bechterev, spondylodiscitis, etc.)
* Presence of a previously diagnosed internal, orthopaedic or neurological disease
* Lateral spinal misalignment caused by a previously diagnosed disease (congenital scoliosis, idiopathic scoliosis, Morbus Scheuermann, etc.)

Exclusion Criteria for non-rowers:

* Active participation in sports associated with an asymmetric load, such as tennis, floorball, hockey and others (training once a week or more)
* Presence of pain caused by a disease for which the person is actively treated (Morbus Bechterev, spondylodiscitis, etc.)
* Presence of a previously diagnosed internal, orthopaedic or neurological disease
* Lateral spinal misalignment caused by a previously diagnosed disease (congenital scoliosis, idiopathic scoliosis, Morbus Scheuermann, etc.)

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Rowers training in the junior and senior category of competitive rowing together with probands from the general population and students of UK FTVS who have never rowed.
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Rotation deviation of the trunk at the level of L3 vertebrae and sway area of COP | one-time measurement
  observation of changed position of the trunk and pelvis
Scoliotic angle in sweep rowers during walking | one-time measurement
  observation of rotational deviation of the trunk during walking
Trunk deviation in the frontal plane and COP deviation | one-time measurement
  observation of later-lateral deviation of he trunk
Magnitude of scoliotic angle | one-time measurement
  observation of the level of scoliotic deviation
Cluster of Laslett testing | one-time measurement
  observation of the mobility of sacroiliac joint

CONTACTS AND LOCATIONS:
Overall Officials: Jitka Malá, PhDr., Study Director — Charles University Prague, Czech Republic
Locations (1):
- Charles University, Faculty of physical education and sport, Prague, Czechia

REFERENCES:
- [Derived] Mikulik L, Mala J, Jajkova K, Opala-Berdzik A. Influence of regularly repeated asymmetric load on the locomotor system in sweep rowers. Sports Biomech. 2024 Dec;23(12):3502-3513. doi: 10.1080/14763141.2024.2382807. Epub 2024 Sep 18. PMID 39295091